CLINICAL TRIAL: NCT03305003
Title: Evaluating How a Mobile App Can Improve Prenatal Care: A Randomized Controlled Trial
Brief Title: Evaluating How a Mobile App Can Improve Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FAM 81-3193
Record Dates: First submitted 2017-09-26; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication modality: spiral notebook (Active Comparator)
  Interventions: Other: Spiral notebook
- Communication modality: mobile application (Experimental)
  Interventions: Other: Mobile application

INTERVENTIONS:
Other: Spiral notebook
  Arms: Communication modality: spiral notebook
Other: Mobile application
  Arms: Communication modality: mobile application

SUMMARY:
Throughout the Military Health System, pregnant mothers are issued a spiral-bound guide that provides week by week information about pregnancy, preventive health messages, appointment information, and space to record their experiences throughout their pregnancy. When used accordingly, the evidence-based guide is an effective tool for motivating patients to participate in their own healthcare and achieve care goals. However, the spiral-bound paper modality results in patients forgetting the book for appointments or losing it. By testing a mobile application (app) from the current publication, the MHS leverages the efforts which created the guide while increasing patient and provider use.

The multisite testing (randomized controlled trial) of a mobile application developed from the current spiral-bound "Pregnancy and Childbirth: A Goal Oriented Guide to Prenatal Care" created by the VA and DoD provides an innovative, cost-effective opportunity to improve provider-patient communication and patient care.

DETAILED DESCRIPTION:
The study was conducted in the women's health and family medicine departments of one community hospital and two medical centers across three states (Georgia, Nevada, and Virginia). In this hospital system, women are distributed a spiral notebook at their obstetric care intake appointment, which generally is scheduled for 8-10 weeks gestation. The spiral notebook is designed for two purposes: 1) patient education of what happens throughout pregnancy, and 2) patient record keeping of the patient's own pregnancy experience, including space for recording weight, blood pressure, and journaling about what they experience between prenatal appointments. The mobile app used in this study was designed for the same two purposes and contained identical content, though through a mobile design interface (available on both Android and iOS platforms). After the pilot study, patient feedback on the mobile app was used to create a beta version. Notable differences were a feature for users to change font size, a search function, and weekly reminders. No substantive content changed. This randomized controlled study had one intervention (mobile application) and one control (standard of care - spiral notebook) group. The study was approved by the first author's Institutional Review Board.

At each medical center, the obstetrics intake nurse serially screened new obstetrics patients for inclusion criteria from May to November 2015. If patients met inclusion criteria, the nurse invited the patient to talk to a research assistant about the study. Exclusion criteria included conditions that would elevate the patient's care to complicated obstetrics care (e.g., cardiovascular disease, diabetes mellitus, renal disorder, etc.). This was intended to capture a low-risk obstetrics patient population that would follow a standard 4-week pathway of care, in which patients attend a prenatal appointment once every four weeks during pregnancy.

The study used pre-assigned block randomization (each block n = 40) to balance the conditions throughout recruitment. Following consent and baseline measures, participants were randomized to the two conditions. Providers were blinded to patient participation in the study.

Surveys were completed at four prenatal appointments, 10-12 weeks, 28 weeks, 32 weeks, and 36 weeks gestation. All data collection was conducted with paper-and-pencil surveys in the clinic, immediately before and following each clinical appointment. At each appointment, patient weight and blood pressure were also recorded from the patient's electronic medical record.

At baseline, self-reported measures included demographics, health literacy, and patient activation. Health literacy was assessed using the self-reported Functional, Communicative, Critical Health Literacy Scale (Ishikawa, Takeuchi, & Yano, 2008) Patient activation was assessed with the validated, licensed patient activation measure (PAM) (Greene & Hibbard, 2012; Greene, Hibbard, Sacks, & Overton, 2013; Hibbard, Mahoney, Stockard, & Tusler, 2005; Hibbard et al., 2004), which uses 13 Likert-type items to create a continuous patient activation measure on a scale of 0 (not activated) to 100 (most activated). PAM was also replicated at time 4 (32 week appointment). As a surrogate measure, patient activation was also assessed at a behavioral level by asking patients at 36 weeks how many mobile apps they had used throughout their pregnancy.

Use was assessed with three measures. Before each appointment, patients completed two items regarding use of the education and engagement tool. First they indicated if they had brought the mobile app/notebook to the appointment with them (yes/no). Then, they reported how frequently they had used the tool over the past month 1) to look for information and 2) to record information (never = 0, once = 1, weekly = 4, or daily = 28).

Following each appointment, patients completed five subscales of the validated Prenatal Interpersonal Processes of Care (PIPC) scale (Wong et al., 2004), including elicitation/responsiveness to the patient, explanations of care, empowerment, patient-centered decision making, and emotional support. Responses to each item were transformed onto a 0 (negative perception) to 100 (positive perception) scale, and items are averaged to create subscales. Then subscales are averaged to calculate the overall PIPC scale.

At delivery, outcomes were recorded from the health record: gestational age, birth weight, and mode of delivery (vaginal or Caesarean section).

ELIGIBILITY:
Inclusion Criteria:

Women (older than 18 years) who initiate obstetrics care (in the Women's Health or Family Health clinics) at the three sites.

Exclusion Criteria:

Exclusion criteria in this study follow the guidelines for patients who are escalated in obstetrical care, to include…

1. Cardiovascular disease
2. Cardiac abnormality
3. Diabetes Mellitus - Type I or Type II
4. Renal disorder
5. Uncontrolled hypertension
6. HIV positive
7. Hepatitis B or C positive
8. History of syphilis/RPR positive
9. Uncontrolled thyroid disease
10. History of previous bariatric surgery
11. Hematologic conditional with the exception of mild anemia
12. Cancer: current or recurrent
13. History of seizure disorder or other neurological condition
14. History of lupus or other autoimmune disorder
15. Antiphospholipid syndrome
16. History of transplant
17. History of genetics disease with known effect on pregnancy
18. Chronic pulmonary disease with the exception of well controlled
19. History of inflammatory bowel disease
20. Thromboembolic disease: current or previous
21. Recurrent pregnancy loss
22. History of isoimmunization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Portability across time | 16-20 weeks gestation, 28 weeks gestation, 32 weeks gestation, 36 weeks gestation
  Question if a patient brings tool to appointments and uses it between appointments
Patient activation across time | 8-10 weeks gestation, 32 weeks gestation
  Patient activation, defined as the knowledge, skills, and confidence to self-manage health
Prenatal Interpersonal Processes of Care across time | 16-20 weeks gestation, 28 weeks gestation, 32 weeks gestation, 36 weeks gestation
  Patient perception of the prenatal providers communicative behavior

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledford CJW, Canzona MR, Cafferty LA, Hodge JA. Mobile application as a prenatal education and engagement tool: A randomized controlled pilot. Patient Educ Couns. 2016 Apr;99(4):578-582. doi: 10.1016/j.pec.2015.11.006. Epub 2015 Nov 10. PMID 26610389
- [Result] Ledford CJW, Womack JJ, Rider HA, Seehusen AB, Conner SJ, Lauters RA, Hodge JA. Unexpected Effects of a System-Distributed Mobile Application in Maternity Care: A Randomized Controlled Trial. Health Educ Behav. 2018 Jun;45(3):323-330. doi: 10.1177/1090198117732110. Epub 2017 Sep 16. PMID 28918669